CLINICAL TRIAL: NCT05422560
Title: Preoperative Embolization of the Inferior Mesenteric Artery in Colorectal Surgery
Acronym: EPAMIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Groupe Hospitalier Mutualiste de Grenoble (Other); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC21.0435
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Embolism Mesenteric
Keywords: Colorectal surgery; Ischemic conditioning; Embolization; Inferior mesenteric artery; Anastomotic fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embolization of the inferior mesenteric artery (Experimental): Only one arm: Patient followed for sigmoid/rectal cancer
  1. Pré-Selection Preoperative consultation, first information to the patient, Validation of IC / NIC, CT-TAP available
  2. Selection Interventional radiology consultation: Consent collection + additional exams
  3. Inclusion V1 - D0:
  4. Follow-up visit V2 - D2: Phone call, pain assessment and analgesic treatments collection
  5. Follow-up visit V3 - D7: Phone call, pain assessment and analgesic treatments collection
  6. Follow-up visit V4 - D21-D30: CT-TAP
  7. Follow-up visit V5 - D30: Digestive surgery consultation + additionnal exams
  8. Surgery V6 - D0: Colic surgery + additional exams
  9. Post-surgery visit V7 - D30: Last visit, additionnal exams
  Interventions: Procedure: Embolization of the inferior mesenteric artery

INTERVENTIONS:
Procedure: Embolization of the inferior mesenteric artery — The procedure is performed in a dedicated angiography room. After local anesthesia, a common femoral arterial approach is performed according to the Seldinger technique with the placement of a 4 French valve introducer.
  Catheterization of the superior mesenteric artery with a Cobra 4F catheter and angiography to confirm patency of the border arcade.
  Catheterization of the inferior mesenteric artery with a 4F cobra/shepherd hook catheter and angiography. Microcatheterization of the artery with a 2.7F or 2.8F microcatheter and embolization with microcoil leaving the first centimeters of the IMA in order not to interfere with the surgery.
  Catheterization of the superior mesenteric artery and final angiography to confirm the reinjection of the inferior mesenteric by the border arcade.
  Removal of the material and manual compression of femoral access. Clinical monitoring for 6 hours and discharge the same day of the procedure.

SUMMARY:
Preoperative embolization of the inferior mesenteric artery in colorectal surgery (EPAMIR).

This is a prospective, monocentric, non-randomized study.

DETAILED DESCRIPTION:
Colorectal surgery accounts for 60,000 acts per year in France. One of the feared complications after colorectal resection surgery is anastomotic leak (5-20% of cases), associated with significant morbidity and mortality. Ischemia of the colorectal or colo-anal anastomosis would be one of the main risk factors for the occurrence of a fistula (REF 1). During the operation, the inferior mesenteric artery is ligated and the remaining colon is vascularized only by Riolan's arch, the link between the networks of the inferior mesenteric artery and the superior mesenteric artery. Arterial ligation by operation is responsible for a transient drop in flow at the level of the anastomosis, while the arch develops.

Preoperative ischemic conditioning by arterial embolization is a technique already used in esophageal surgery (REF 2). The objective is to embolize the arterial branches that will be ligated during surgery a few weeks before the resection procedure, in order to allow hypertrophy of the remaining branches to allow better vascularization of the anastomosis on the day of the intervention. The CHUGA is one of the motor centers of this technique. In our experience, embolization performed 3 to 4 weeks before esophageal surgery allows a reduction in the rate of fistulas (p=0.02). These results made it possible to aggregate other centers towards this technique, and a request for PHRC-K is in progress.

In the context of ischemic conditioning before colorectal surgery, a proof of concept on 5 patients has just been completed by the University Hospital of Nîmes (REF 3) of which Dr Ghelfi (Radiologist) and Dr Trilling (Colorectal Surgeon) are investigators. The preliminary results seem suggested.

The responsibility and safety of preoperative embolization of the inferior mesenteric artery have already been validated by meta-analyses of data from patients who received AMI embolization before placement of a covered aortic stent (REF 4).

The objective of this study is to show that ischemic conditioning improves the vascular supply of the colon for risky procedures in colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patient to benefit from left colonic surgery or rectal surgery with upper ligation of the inferior mesenteric artery and colorectal or colo anastomosis
* Person affiliated to or benefiting from social security
* Person who has given written informed consent

Exclusion Criteria:

* History of digestive resection or abdominal aorta surgery
* Renal failure with GFR < 30 ml/min (MDRD)
* History of severe allergy to iodine contrast medium
* Pregnant, parturient, lactating women
* Patient subject to a legal protection measure or unable to express his non-opposition (guardianship, curatorship)
* Patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Measure of the Riolan arch (diameter in mm) | CT-TAP before embolization and CT-TAP between 3 and 4 weeks after embolization, before surgery.
  Evaluation of the difference in size (diameter in mm) of the Riolan arch

SECONDARY OUTCOMES:
Evaluation of the rate of complications related to preoperative embolization of the inferior mesenteric artery | Between 21 and 30 days after embolization, before surgery.
  Pain assessment, analgesic treatments collection, diarrhea, blood in the stool, hypertermia, Hematoma at the puncture site, occurence of adverse events.
Evaluation of the rate of anastomotic fistulas after colo-rectal surgery | 30 days after colorectal surgery
  CT-TAP, occurence of adverse events.
Evaluation of the rate of complications related to colorectal surgery | 30 days after colorectal surgery
  CT-TAP, occurence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Julien GHELFI, MD, Principal Investigator — Grenoble Alpes University Hospital
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Groupe Hospitalier Mutualiste, Grenoble
  - Grenoble Alpes University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] van der Pas MH, Haglind E, Cuesta MA, Furst A, Lacy AM, Hop WC, Bonjer HJ; COlorectal cancer Laparoscopic or Open Resection II (COLOR II) Study Group. Laparoscopic versus open surgery for rectal cancer (COLOR II): short-term outcomes of a randomised, phase 3 trial. Lancet Oncol. 2013 Mar;14(3):210-8. doi: 10.1016/S1470-2045(13)70016-0. Epub 2013 Feb 6. PMID 23395398
- [Background] Snijders HS, Wouters MW, van Leersum NJ, Kolfschoten NE, Henneman D, de Vries AC, Tollenaar RA, Bonsing BA. Meta-analysis of the risk for anastomotic leakage, the postoperative mortality caused by leakage in relation to the overall postoperative mortality. Eur J Surg Oncol. 2012 Nov;38(11):1013-9. doi: 10.1016/j.ejso.2012.07.111. Epub 2012 Sep 3. PMID 22954525
- [Background] Posma LA, Bleichrodt RP, van Goor H, Hendriks T. Transient profound mesenteric ischemia strongly affects the strength of intestinal anastomoses in the rat. Dis Colon Rectum. 2007 Jul;50(7):1070-9. doi: 10.1007/s10350-006-0822-9. PMID 17205202
- [Background] Ghelfi J, Brichon PY, Frandon J, Boussat B, Bricault I, Ferretti G, Guigard S, Sengel C. Ischemic Gastric Conditioning by Preoperative Arterial Embolization Before Oncologic Esophagectomy: A Single-Center Experience. Cardiovasc Intervent Radiol. 2017 May;40(5):712-720. doi: 10.1007/s00270-016-1556-2. Epub 2017 Jan 3. PMID 28050659
- [Background] Manunga JM, Cragg A, Garberich R, Urbach JA, Skeik N, Alexander J, Titus J, Stephenson E, Alden P, Sullivan TM. Preoperative Inferior Mesenteric Artery Embolization: A Valid Method to Reduce the Rate of Type II Endoleak after EVAR? Ann Vasc Surg. 2017 Feb;39:40-47. doi: 10.1016/j.avsg.2016.05.106. Epub 2016 Aug 12. PMID 27531083